CLINICAL TRIAL: NCT07399015
Title: Intermediate-size Expanded Access Protocol (EAP): Mifomelatide for the Treatment of Cachexia in Adults With Advanced, Unresectable PDAC
Brief Title: Expanded Access to Mifomelatide for Cachexia in Adults With Advanced PDAC
Status: Available | Type: Expanded Access
Sponsor: Endevica Bio (Industry)
Collaborators: Kalohexis (Industry)
Responsible Party: Sponsor
Other Study IDs: Mifomelatide-EAP-01
Record Dates: First submitted 2026-01-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma (mPDAC); Unresectable Pancreatic Ductal Adenocarcinoma; Metastatic PDAC
Keywords: cancer weight loss; advanced pancreatic cancer; metastatic pancreatic cancer; cancer cachexia; advanced pancreatic ductal adenocarcinoma; weight loss in pancreatic cancer
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia; Pancreatic Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: mifomelatide — Eligible participants will receive 25 mg mifomelatide daily by subcutaneous (SC) injection for up to 13 weeks.

SUMMARY:
An expanded access program (EAP) allows doctors to give medicine to seriously ill patients before it is approved by local regulatory agencies.

The goal of this Expanded Access Protocol is to provide access to mifomelatide for eligible cachectic adult patients with advanced, unresectable pancreatic ductal adenocarcinoma (PDAC) who lack satisfactory therapeutic alternatives for their cancer cachexia and are not eligible for current mifomelatide clinical trials.

A participant may receive mifomelatide under this EAP if:

* A licensed doctor submits a request,
* The participant is eligible
* The country allows the EAP

DETAILED DESCRIPTION:
This is an expanded access program (EAP) providing access to mifomelatide for participants with advanced, unresectable pancreatic ductal adenocarcinoma (PDAC) and cachexia, prior to approval by local regulatory agencies.

Availability of the EAP is dependent upon physician request, country eligibility and local/country regulations. Physicians may request access to the EAP for participants who they feel may benefit from mifomelatide and meet the eligibility criteria.

Once enrolled, participants will receive mifomelatide by subcutaneous injection once daily for up to 13 weeks.

Participants will be asked to follow the standard of care treatment for their cancer as outlined by their treating physician. Participants will be followed for safety up to 30 days after their final treatment. Physicians will be required to report safety data to Kalohexis (a spin off company from Endevica Bio).

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age
2. Documented histologic or cytologic diagnosis of advanced, unresectable PDAC
3. Current cachexia (documented in medical records) as defined by Fearon criteria based on at least one of the following three weight loss conditions in the 6 months prior to enrollment:

   1. Weight loss of at least 5%
   2. Weight loss of at least 2% together with a BMI <20 kg/m2 and/or
   3. Weight loss of at least 2% together with sarcopenia
4. Eastern Cooperative Oncology Group (ECOG) status of ≤ 3 and life expectancy ≥ 4 months
5. Lack of satisfactory therapeutic alternatives for their cancer cachexia
6. Willing and able to safely self-inject or be injected by a caregiver daily
7. Not eligible to participate in ongoing clinical trials of the investigational drug
8. Willing and able to sign informed consent

Exclusion Criteria:

1. Patients with BMI > 35
2. Known hypersensitivity to mifomelatide or its formulation
3. Significant medical conditions or illnesses that might increase the risk-benefit ratio of participating in this EAP as determined by the

   Treating Physician, which may include:
   * Patients with swallowing abnormalities, malabsorption syndromes, severe short or inflammatory bowel syndromes, or other conditions that in the Treating Physician's opinion could impair food consumption or metabolism
   * Receiving exclusive tube feeding or parenteral nutrition at the time of enrollment
   * History of weight loss surgery including gastric stapling, or bypass
   * ANC < 1.5 x 109/L
   * AST and/or ALT > 3 x ULN (> 5 x ULN in the presence of documented liver metastases)
   * Total bilirubin > 1.5 x ULN (> 3 x ULN in the presence of documented Gilbert's Syndrome)
   * Creatinine clearance calculated by Cockcroft and Gault equation < 50 mL/min Uncontrolled diabetes defined as HbA1c >7%
4. Currently pregnant, breastfeeding or planning to become pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dan Marks, MD, PhD, Study Director — Endevica Bio